CLINICAL TRIAL: NCT05109598
Title: A Clinical Trial Comparing the Immunogenicity of Recombinant New Coronavirus Vaccine (CHO Cells) Among People Aged 3 to 17 and 18 to 59 Years of Age.
Brief Title: Clinical Trial of Immunogenicity Bridging of a Recombinant New Coronavirus（COVID-19） Vaccine (CHO Cell)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anhui Zhifei Longcom Biologic Pharmacy Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LKM-2021-NCV03
Record Dates: First submitted 2021-11-04; First posted 2021-11-05 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: COVID-19
Keywords: Recombinant Novel Coronavirus Vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Population I (Experimental): Population I has 400 subjects aged 3 to 17 who were recruited by this trial.
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cell)
- Population II (Experimental): Population II will use 400 subjects aged of 18-59 in the phase III clinical trial in China whose blood has been collected.
  Interventions: Biological: Recombinant new coronavirus vaccine (CHO cell)

INTERVENTIONS:
Biological: Recombinant new coronavirus vaccine (CHO cell) — Intramuscular injection of deltoid muscle of upper arm of 25μg/0.5ml/person /dose Recombinant new coronavirus vaccine (CHO cells).

SUMMARY:
Popular topic: A clinical trial comparing the immunogenicity of recombinant New Coronavirus vaccine (CHO cells) among people aged 3 to 17 and 18 to 59 years of age.

Overall design:Non inferiority test design was used to evaluate the immunogenicity of the vaccine inoculated to the age group of 3~17 and the age of 18~59. The non inferiority hypothesis test was conducted with the results of immunogenicity of the 18-59 year old group in China in the phase III clinical trial of recombinant New Coronavirus vaccine (CHO cell).

Study population:400 healthy people aged 3 to 17 years old, both male and female.

DETAILED DESCRIPTION:
Study population:A total of 400 healthy people aged 3 ~ 17 were enrolled (including 130 cases aged 3 ~ 5, 150 cases aged 6 ~ 11, and 120 cases aged 12 ~ 17)，both male and female.

Overall design:Non inferiority test design was used to evaluate the immunogenicity of the vaccine inoculated to the age group of 3~17 and the age of 18~59. The non inferiority hypothesis test was conducted with the results of immunogenicity of the 18-59 year old group in China in the phase III clinical trial of recombinant New Coronavirus vaccine (CHO cell).

Immunization program: Three doses were inoculated in 0, 1 and 2 months. Dose:25μg/0.5mL/dose.

Safety endpoint:

1. AE and SAE:Collect all adverse events (AES) 30 minutes after each dose of vaccination, all AES 0-7 days (including solicited and non solicited AES), all AES 8-30 days (non solicited AES), and all SAE from the first dose of vaccination to 12 months after the whole course of immunization.
2. Vital signs and physical examination:

   All subjects underwent axillary temperature examination every day during the screening period, before the next dose of vaccination and within 7 days after each dose of vaccination.

   All subjects underwent physical examination (skin and cardiopulmonary auscultation) during the screening period.
3. Pregnancy events:

   For women of childbearing age, urine pregnancy test should be carried out before each dose of vaccination.

   The pregnancy events occurred within 12 months from the first dose of vaccine to the whole course of immunization were collected.
4. ADE / VED risk monitoring:

After vaccination (at least one dose of test vaccine) (at each visit), remind the subjects to contact the investigator in time for fever and / or respiratory symptoms (such as dyspnea, sore throat, etc.) and covid-19 suspected or confirmed cases during the study. If the subject is suspected or confirmed to be infected with sars-cov-2 during the test, he must go to the local Xinguan designated hospital for hospitalization diagnosis and treatment. Detailed case investigation shall be conducted for confirmed cases. In case of severe or dead cases of new crown infection, an expert meeting shall be held to conduct special investigation and evaluate whether it is ADE/ VED.

ELIGIBILITY:
Inclusion Criteria:

1. At least 3 ~ 17 years old (both included);
2. The subject voluntarily agrees to participate in the study, and / or the guardian of the subject voluntarily agrees to the child to participate in the study. The subject himself (8-17 years old) and the guardian sign the informed consent form, and can provide valid identity certificates to understand and comply with the requirements of the test protocol;
3. The subject and / or the guardian of the subject have the ability to understand (non illiterate) the research procedures and promise to participate in regular follow-up according to the research requirements;
4. There is no high or medium risk area, overseas travel history or residence history in the past 14 days; In the past 14 days, no confirmed case of New Coronavirus infection, asymptomatic infection or suspected cases had been found. And there was no contact history of patients with fever or respiratory symptoms from high and medium risk areas in the past 14 days; Personnel in non isolation period;
5. Male and female subjects with fertility agreed to take effective contraceptive measures from the beginning of the study to 2 months after the whole vaccination.

Exclusion Criteria:

1. The results of physical examination during screening period are abnormal and clinically significant (not suitable for vaccination) as determined by clinicians;
2. Suspected or confirmed fever within 72 hours before enrollment (including the day of enrollment) (> 14 years old, axillary temperature ≥ 37.3 ℃; ≤ 14 years old, axillary temperature ≥ 37.5 ℃);
3. Have a history of severe allergy to any component of the test vaccine, including aluminum preparation, such as anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, dyspnea, angioneurotic edema, etc; Or have a history of the above serious side effects after the use of any vaccine or drug in the past;
4. had previous history of SARS and SARS-CoV-2.
5. Taking antipyretics or painkillers within 24 hours before the first dose of vaccine;
6. persons who have been vaccinated with New Coronavirus or inoculated with live attenuated vaccine within 7 days or within 7 days before the first dose of vaccine are inoculated with inward subunit vaccine and / or inactivated vaccine.
7. Have received blood or blood related products, including immunoglobulin, within 3 months before the vaccination of the test vaccine; Or planned use during the study;
8. Persons suffering from the following diseases:

   ① Digestive system diseases (such as diarrhea, abdominal pain, vomiting, etc.) in the past 7 days;

   ② Suffering from congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc;

   ③ History of congenital or acquired immune deficiency or autoimmune diseases or receiving immunomodulator treatment within 6 months, such as immunosuppressive dose of Glucocorticoid (dose reference: equivalent to prednisone 20mg / day, more than one week); Or monoclonal antibody; Or thymosin; Or interferon, etc; However, topical medication (such as ointment, eye drops, inhalants or nasal sprays) is allowed;

   ④ It is known that it is diagnosed with infectious diseases, such as active tuberculosis, viral hepatitis present, human immunodeficiency virus infection or Treponema pallidum infection.

   ⑤ Neurological diseases or neurodysplasia (e.g., convulsions, migraines, epilepsy, stroke, seizures in the last three years, encephalopathy, focal neurological deficit, Guillain Barre syndrome, encephalomyelitis or transverse myelitis); History of psychosis or family history;

   ⑥ Functional absence of spleen, and absence of spleen or splenectomy for any reason;

   ⑦ There are serious chronic diseases or disease in progress can not be controlled smoothly, such as diabetes, drugs can not control hypertension.

   ⑧ Severe liver and kidney diseases; Respiratory diseases that currently require daily drug treatment (e.g., chronic obstructive pulmonary disease [COPD], asthma) or any treatment for aggravation of respiratory diseases (e.g., aggravation of asthma) in the last 5 years; A history of serious cardiovascular disease (such as congestive heart failure, cardiomyopathy, ischemic heart disease, arrhythmia, conduction block, myocardial infarction, cor pulmonale) or myocarditis or pericarditis;

   ⑨ Thrombocytopenia, any coagulation dysfunction or anticoagulant treatment;

   ⑩ Cancer patients (except basal cell carcinoma);
9. Lactating women or pregnant women (including women of childbearing age with positive urine pregnancy test), or women or their partners who have pregnancy plans within 2 months after the whole vaccination of the test vaccine;
10. Those who have participated or are participating in other clinical trials, and the relevant visits have not been completed, or are clearly vaccinated after the completion of the new crown vaccine;
11. The researcher believes that the subject has any disease or condition that may put the subject at unacceptable risk; The subjects were unable to meet the protocol requirements; Interference with the evaluation of vaccine response.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
Immunogenic end point | 14 days after full vaccination
  The positive rate of sars-cov-2 neutralizing antibody, RBD protein binding antibody (IgG) GMT and 14 days after the whole course immunization of the test vaccine in the target population.
The number of adverse events after intramuscular injection | from the first dose to 1 month after the whole course of immunization
  All adverse events (AE) from the first dose to 1 month after the whole course of immunization
The number of serious adverse events after intramuscular injection | from the first dose to 12 months after the whole course of vaccination.
  Incidence of all serious adverse events (SAE) and vaccine related SAE from the first dose to 12 months after the whole course of vaccination.

SECONDARY OUTCOMES:
Immunopersistence results | 6 months after the last dose of vaccination
  The positive rate of sars-cov-2 neutralizing antibody, RBD protein binding antibody (IgG) GMT and 6 months after the whole course immunization of the test vaccine in the target population.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Huang, Study Director — Hunan Provincial Center for Disease Control and Prevention
Locations (1):
- Hunan Provincial Center for Disease Control and Prevention, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gao L, Li Y, He P, Chen Z, Yang H, Li F, Zhang S, Wang D, Wang G, Yang S, Gong L, Ding F, Ling M, Wang X, Ci L, Dai L, Gao GF, Huang T, Hu Z, Ying Z, Sun J, Zuo X. Safety and immunogenicity of a protein subunit COVID-19 vaccine (ZF2001) in healthy children and adolescents aged 3-17 years in China: a randomised, double-blind, placebo-controlled, phase 1 trial and an open-label, non-randomised, non-inferiority, phase 2 trial. Lancet Child Adolesc Health. 2023 Apr;7(4):269-279. doi: 10.1016/S2352-4642(22)00376-5. Epub 2023 Feb 17. PMID 36803632